CLINICAL TRIAL: NCT00733941
Title: Interval Training: Training, Detraining and Retraining; an Interventional Study
Brief Title: Interval Training in Young Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4.2008.1755
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Healthy Subjects; Exercise Test
Keywords: Exercise test; Running; Arterial diameter; Monitoring, physiologic; Oxygen Consumption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High frequency training (Experimental): 24 interval exercises performed 8 times per week
  Interventions: Behavioral: High frequency training
- Normal frequency training (Experimental): 24 interval exercises performed 3 times per week
  Interventions: Behavioral: normal frequence training

INTERVENTIONS:
Behavioral: High frequency training — 24 training sessions, 8x weekly, followed by detraining phase 8 weeks, and retraining
  Arms: High frequency training
Behavioral: normal frequence training — 24 training sessions, 3x weekly, followed by detraining phase 8 weeks, and retraining
  Arms: Normal frequency training

SUMMARY:
Individuals who participate in regular physical exercise possess a lower prevalence of cardiovascular risk factors such as hypertension, type 2 diabetes, obesity and hypercholesterolemia, and aerobic exercise is therefore considered an important adjuvant therapy in risk factor modification and to promote health.

The main focus of the present study is therefore to detect how rapid it is possible to increase aerobic capacity with interval running exercise.

The hypothesis is that it is possible to improve maximal oxygen uptake faster when increasing training frequency. The total gain in maximal oxygen uptake will however be the same between the two groups when they have performed the same amount of training

DETAILED DESCRIPTION:
We will perform aerobic interval training at an intensity of 90-95% of maximum heart rate in healthy individuals. The subjects will be randomly assigned to carry out a total of 24 exercise-sessions, either at 3 times per week or 8 times per week.

The two groups will carry out 24 training sessions before 8 weeks of detraining will provide how rapidly aerobic capacity is lost due to inactivity. After the detraining period a retraining phase is introduced to detect if improvements in aerobic capacity occur more rapidly compared to before the first training period

The subjects will be tested for oxygen uptake, pumping capacity of the heart, blood volume, skeletal muscle enzyme activity, endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* BMI<27, non-smokers, train less that 1-2 times per week, VO2max <60 for male and <50 for female.

Exclusion Criteria:

* Hypertension, diabetes and cardiovascular disease.

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Oxygen uptake | Before and after the training-, detraining- and retraining-phase

SECONDARY OUTCOMES:
Cardiac function and skeletal muscle enzyme activity | After training, detraining and retraining

CONTACTS AND LOCATIONS:
Overall Officials: Øivind Rognmo, PhD, Principal Investigator — Norwegian University of Science and Technology; Ulrik Wisløff, Professor, Principal Investigator — National Taiwan Normal University
Locations (2):
- Norway (2):
  - Norwegian University of Science and Technology, Trondheim
  - NTNU, Trondheim

REFERENCES:
- [Result] Hatle H, Stobakk PK, Molmen HE, Bronstad E, Tjonna AE, Steinshamn S, Skogvoll E, Wisloff U, Ingul CB, Rognmo O. Effect of 24 sessions of high-intensity aerobic interval training carried out at either high or moderate frequency, a randomized trial. PLoS One. 2014 Feb 7;9(2):e88375. doi: 10.1371/journal.pone.0088375. eCollection 2014. PMID 24516645